CLINICAL TRIAL: NCT05980611
Title: Evaluation of Nasal IL 1 Beta ,IL 3 Level and Their Effects on Disease Severity in COPD
Brief Title: Nasal IL 1 Beta ,IL 3 Level and Their Effects in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermen Abuelkassem, lecturer, Assiut University
Other Study IDs: nasal IL B,IL 3 ,COPD
Record Dates: First submitted 2023-07-05; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Copd Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- copd patients with high upper airway symptoms: The SNOT22 nasal subdomain (SNOT22nasal) consists of seven questions (no. 1-5 + 7-8), which include: "need to blow nose", "sneezing", "runny nose", "nasal obstruction", "loss of smell or taste", "post-nasal discharge" and "thick nasal discharge". the total SNOT22 has been found to have a median score of 7 points in healthy volunteers
  Interventions: Diagnostic Test: IL B,IL 3 in nasal swap and serum
- copd patients with low upper airway symptoms: The SNOT22 nasal subdomain (SNOT22nasal) consists of seven questions (no. 1-5 + 7-8), which include: "need to blow nose", "sneezing", "runny nose", "nasal obstruction", "loss of smell or taste", "post-nasal discharge" and "thick nasal discharge". the total SNOT22 has been found to have a median score of 7 points in healthy volunteers
  Interventions: Diagnostic Test: IL B,IL 3 in nasal swap and serum

INTERVENTIONS:
Diagnostic Test: IL B,IL 3 in nasal swap and serum — Interleukin (IL)-1-beta and IL-3 will be measured in patients' serum and supernatant from the nasal swap using enzyme linked immunosorbent assay (ELISA).

SUMMARY:
Chronic obstructive pulmonary disease is associated with systemic and local inflammation. exposure to harmful gases and particles play important role in initiating the inflammatory processes leading to the development of COPD. In high- and medium-income countries, tobacco smoking is considered the predominant source of these noxious elements.1 Asthma, COPD, rhinitis and rhinosinusitis (RS) are chronic diseases of the respiratory tract with an estimated global prevalence of about 12%.2The concept of united airways diseases (UAD) was formulated on the initial observation of the coexistence of allergic rhinitis and chronic rhinosinusitis with asthma.3

DETAILED DESCRIPTION:
. COPD patients asscioted with upper airway disease either high symptoms or low symptoms according to The 22-item Sino Nasal Outcome Test .Data will be collected through: History and examination of the upper airways and COPD symptomatology. History of smoking, medication, admission and acute exacerbation . Pulmonary function tests to confirm diagnosis and degree of obstruction. Diagnosis of COPD will be confirmed by the presence of irreversible airflow obstruction, post-bronchodilator FEV1/FVC ratio of less than 0.7. Severity of airflow obstruction will be graded according to the GOLD criteria [9] using CAT questionnaire to assess degree of COPD burden.[10] The 22-item Sino Nasal Outcome Test (SNOT22) will assess chronic rhinosinusitis symptoms and includes nasal and more general symptoms such as fatigue [11]. Each symptom is scored from 0 (no symptoms) to 5 (symptoms as bad as they can be"). The maximum score is 110, with an MCID of 9 points [12].

The SNOT22 nasal subdomain (SNOT22nasal) consists of seven questions (no. 1-5 + 7-8), which include: "need to blow nose", "sneezing", "runny nose", "nasal obstruction", "loss of smell or taste", "post-nasal discharge" and "thick nasal discharge". A cut-off for normality (or MCID) has been not validated, however the total SNOT22 has been found to have a median score of 7 points in healthy volunteers [12] Clinical markers in COPD symptom severity: Dyspnea will be graded using the mMRC 5-point scale.13 Physical Activity The 6MWD will be measured in accordance with the standard protocol with modifications.14 The latter were a shorter walking lap of 50 m instead of 60 m . Participants rested for 10 min before the test and then followed a straight corridor with a length of 25 m which was marked every 5 m. The turnaround points were set up with a red cone, and the distance walked in 6 minutes was recorded. Standardized phrases of encouragement were given during the test. Disease-specific HRQoL for COPD was measured by the CAT and the SGRQ questionnaires. The range of the total score is from 0 to 40 for the former and from 0 to 100 for the latter questionnaire, and high scores are indicative of poorer HRQoL

ELIGIBILITY:
Inclusion Criteria:We included patients according to the following inclusion criteria:

* age ≥ 40 years
* History of smoking > ten pack-years of tobacco
* Post- bronchodilator Forced Expiratory Volume 1 s (FEV1)/Forced Vital Capacity (FVC) index <0.70.

Exclusion Criteria:self-reported or physician- diagnosed asthma and reversibility for beta 2 agonist above 400 ml and 15% from baseline FEV1

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: copd patients
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
degree of Upper Airway inflammation and severity of COPD | 1 year
  patients with high UAD mostly affect degree of obstruction which assessed by FEV1 in PFT

SECONDARY OUTCOMES:
high UAD and severity of COPD togeher and impact on quality of life in those patients | 1 year
  patients with copd and nasal involvement and quality of life by using saint george questionnaire

IPD SHARING:
Plan to Share IPD: Undecided